CLINICAL TRIAL: NCT02502669
Title: A Double-Blind, Randomized, Placebo-Controlled Dose-Ranging Study Evaluating the Efficacy and Safety of Once Weekly High Dose Oral Finasteride in the Treatment of Severe Nodulocystic Acne
Brief Title: Finasteride Treatment of Severe Nodulocystic Acne
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Elorac, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EL-1006-01-01
Record Dates: First submitted 2015-07-10; First posted 2015-07-20 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: NODULOCYSTIC ACNE
Keywords: acne; nodulocystic; finasteride; 5 alpha reductase inhibitor
MeSH Terms: conditions — Acne Vulgaris | interventions — Finasteride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Finasteride 23.5 mg tablets group (Active Comparator): Finasteride 23.5mg tablets and large placebo tablets once per week
  Interventions: Drug: Finasteride 23.5 mg tablets; Drug: Placebo tablets
- Finasteride 33.5 mg tablets group (Active Comparator): Finasteride 33.5 mg tablets and small placebo tablets once per week
  Interventions: Drug: Finasteride 33.5 mg tablets; Drug: Placebo tablets
- Placebo group (Placebo Comparator): Large and small placebo tablets once per week
  Interventions: Drug: Placebo tablets

INTERVENTIONS:
Drug: Finasteride 23.5 mg tablets
  Arms: Finasteride 23.5 mg tablets group
Drug: Finasteride 33.5 mg tablets
  Arms: Finasteride 33.5 mg tablets group
Drug: Placebo tablets

SUMMARY:
Double-blind, randomized, placebo-controlled, dose-ranging study to evaluate the efficacy and safety of once weekly, high dose oral finasteride compared to placebo for the treatment of severe nodulocystic acne in male subjects.

DETAILED DESCRIPTION:
There will be 180 male subjects in this study. The study is composed of a Screening Period of up to 30 days during which inclusion / exclusion criteria will be reviewed, screening laboratory results will be obtained and medication washouts will be done as required. Subjects will complete the sexual function questionnaire and depression scale. A one day Baseline Period (Day 0), during which baseline assessments of acne lesion counts, physical examination and Investigator's Global Assessment Scale will be done. The Baseline Period will be followed by a 12-week randomized double-blind Treatment Period, in which subjects will be randomized into Finasteride 23.5 mg group, 33.5 mg group, or placebo group. During the Treatment Period, subjects will visit the study site Day 14, Day 28, and Day 56 for acne lesion counts and review of diaries, concomitant medications and adverse events. On Day 84 subjects will return to clinic for acne lesion counts and review of diaries, concomitant medications, adverse events and remaining study drug will be counted and collected. A physical exam and vital signs, Investigator Global Assessment, Subject Assessment of Efficacy, depression scale and sexual function questionnaire will be completed before the subject is discharged from the study.

ELIGIBILITY:
Inclusion Criteria:

1. Subject voluntarily agrees to participate in this study and signs an IRB-approved informed consent prior to performing any of the screening procedures.
2. Males 18 years to 35 years of age.
3. Except for severe nodulocystic acne, subject is in generally good health.
4. Ten (10) or more nodular lesions (facial and/or truncal).
5. Weight between 40 and 110 kg.
6. No significant disease or clinically significant finding in a physical examination.
7. No clinically significant abnormal laboratory value.
8. No clinically significant abnormal vital sign measurement.
9. Subject is able to swallow pills.
10. Subject agrees to use a medically acceptable form of barrier-method contraception (e.g. condoms with spermicide or abstinence).
11. Subject is willing and able to cooperate to the extent required by the protocol.

Exclusion Criteria:

1. Female subjects will be excluded from the study.
2. Subject with acne conglobata, acne fulminans, secondary acne (chloracne, drug-induced acne, etc.), pyoderma faciale, sinus tracks.
3. Subject with a wash out period from Baseline for topical treatment on the skin less than: Corticosteroids, antibiotics, antibacterials, antiseptics, retinoids, other anti-inflammatory drugs or other acne treatment (2 weeks); Cosmetic procedures (1 week); Photodynamic therapy and laser therapy for acne (3 months).
4. Subject with a washout period from Baseline for systemic treatment less than: Corticosteroids, antibiotics (4 weeks), spironolactone (3 months), other systemic acne treatments (6 months), cyproterone acetate (6 months), lithium, anticonvulsants, barbiturates, androgenic and anabolic steroids, testosterone, estrogen, anti-tuberculous drugs, cyclosporine, and azathioprine (6 months), surgical treatment of acne (12 months), finasteride or other 5α-reductase inhibitors (12 months). (Table 2)
5. Subjects with current or history of prostatic disease including benign prostatic hypertrophy, or surgery on prostate.
6. Known history or presence of any clinically significant unstable medical condition(s) which in the opinion of the investigator could pose a risk for the safety of the subject, e.g. diabetes, cardiovascular, liver or kidney disease.
7. Subjects with any skin disease or other condition that might interfere with the evaluation of nodular acne.
8. Known history or suspected carcinoma.
9. Allergy to finasteride or any other ingredients in the study medications.
10. Subjects with history in past 12 months of active addiction, abuse, misuse and/or dependence on drugs or alcohol.
11. Use of investigational drug within 90 days prior to Day 1

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 106 (Actual)
Dates: Start 2015-07; Primary Completion 2017-06-06 (Actual); Study Completion 2017-06-06 (Actual)

PRIMARY OUTCOMES:
Acne Nodular Lesion Count | 12 Weeks
  Change from Baseline to week 12 in the total number of nodular lesions

SECONDARY OUTCOMES:
Proportion of Subjects who achieve at least a 75% reduction in total number of nodular lesions | 12 Weeks
  Change from Baseline to week 12 in the total number of nodular lesions
Investigator's Global Assessment Scale of Acne Severity | 12 Weeks
  Change from Baseline to week 12
Non-Inferiority (NI) for non-nodulocystic inflammatory lesions | 12 Weeks
  The NI bound will be larger of 10% reduction or a count of 4 lesions.
Change in total number of nodular lesions. | 2, 4, and 8 weeks
  Change from baseline to weeks 2, 4 and 8.
Proportion of subjects with 2 category improvement on Investigator's Global Assessment Scale | 12 Weeks
  Change from Baseline to week 12

CONTACTS AND LOCATIONS:
Overall Officials: Scott B. Phillips, MD, Study Director — Elorac, Inc.
Locations (25):
- United States (25):
  - Omni Dermatology, Inc., Phoenix, Arizona
  - Burke Pharmaceutical Research, Hot Springs, Arkansas
  - Dr. Ronald Moy, Beverly Hills, California
  - Axis Clinical Trials, Los Angeles, California
  - Orange County Research Center, Tustin, California
  - Horizons Clinical Research Center, LLC., Denver, Colorado
  - MOORE Clinical Research, Inc., Brandon, Florida
  - Advanced Medcial Research Institiute, Miami Lakes, Florida
  - Park Avenue Dermatology, Orange Park, Florida
  - International Clinical Research, Sanford, Florida
  - Lenus Research & Medical Group, Sweetwater, Florida
  - Marietta Dermatology Clinical Research, Inc., Marietta, Georgia
  - MedaPhase, Inc., Newnan, Georgia
  - Northwest Clinical Trials, Boise, Idaho
  - Glazer Dermatology, Buffalo Grove, Illinois
  - Northwestern University, Chicago, Illinois
  - Summit Dermatology, Oakbrook Terrace, Illinois
  - Dawes Fretzin Clinical Research Group. LLC, Indianapolis, Indiana
  - The Indiana Clinical Trials Center, PC, Plainfield, Indiana
  - Hamzavi Dermatology, Fort Gratiot, Michigan
  - MediSearch Clinical Trials, Saint Joseph, Missouri
  - Greenwich Village Dermatology, New York, New York
  - UHCMC Skin Study Center, Cleveland, Ohio
  - Paddington Testing Co., Inc., Philadelphia, Pennsylvania
  - Invocare Clinical Research Center, West Columbia, South Carolina